CLINICAL TRIAL: NCT06227026
Title: Pilot Study of Anti-CD19 Chimeric Antigen Receptor T Cells (CAR-T Cells) for the Treatment of Relapsed/Refractory CD19+ Malignancies
Acronym: PRODIGY
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI143560
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Masking Description: This study will utilize a staggered enrollment design. Following the CAR-T infusion of the first subject, further enrollment will be paused for a 28 day safety observation period. If deemed safe by the Data Safety Monitoring Committee (DSMC) after this period (i.e. no stopping rules have been satisfied), enrollment of the second subject may proceed. Following the CAR-T infusion of the second subject, enrollment will again be paused for a 28 day safety observation period. Enrollment of the remaining subjects may only proceed after approval from the DSMC following the safety observation period for the second subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Anti-CD19 CAR-T Cell Infusion (Experimental)
  Interventions: Biological: Anti-CD19 CAR-T cells

INTERVENTIONS:
Biological: Anti-CD19 CAR-T cells — Anti-CD19 CAR-T cells are autologous T cells, engineered to express an extracellular single chain variable fragment (scFv) derived from a murine anti-human CD19 hybridoma clone FMC63 linked in frame to hinge region derived from human CD8, transmembrane domain derived from Tumor Necrosis Factor Receptor Super Family 19 (TNFRSF19) the transactivation costimulatory domain 4-1BB, and CD3 zeta signaling domain (Miltenyi Biotec Inc). Anti-CD19 CAR-T cells will be cryopreserved in infusible cryomedia for a later infusion. Anti-CD19 CAR-T cells will be administered in 1 to 3 bags. Bag aliquoting, cell content and cryomedia composition will be done according to specifications in the CMC.

SUMMARY:
This is an open label, non-randomized, phase 1 study of anti-CD19 CAR-T cells against relapsed CD19 positive NHL, CLL and ALL based in a lymphodepletion regimen (fludarabine and cyclophosphamide) and using a CellReGen-based process for manufacturing CAR-T cells.

This study will utilize a staggered enrollment design with a safety observation period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 years.
* Histologically confirmed relapsed or refractory CD-19+ malignancy, including: non-Hodgkin lymphoma (NHL), acute lymphoblastic leukemia (ALL), Chronic Lymphocytic Leukemia (CLL)/Richter's syndrome. CD-19+ must be confirmed by immunohistochemistry or flow cytometry analysis.
* Subjects who have relapsed or refractory disease after failing at least 2 or more prior lines of therapy.
* ECOG Performance Status ≤ 2.
* Life expectancy > 12 weeks.
* Willing to consent to 15 years of follow-up as part of IRB 110692: Long-Term Evaluation of the Biology and Outcomes of Hematopoietic Stem Cell Transplantation
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count (ANC) ≥ 500/mm3
    * Platelet count ≥ 10,000/mm3
    * Hemoglobin ≥ 8 g/dL
  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN).
    * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
  * Renal:

    * Serum Creatinine ≤ 2 x institutional upper limit of normal (ULN) or eGFR >30 ml/min/1.73m2
* For subjects of childbearing potential: Negative pregnancy test or evidence of post-menopausal status or evidence of permanent surgical sterilization. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Subjects < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
  * Subjects ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago
* Subjects of childbearing potential and subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception as described in Section 5.4.1.
* Recovery to baseline or ≤ Grade 2 CTCAE v5.0 from toxicities related to any prior cancer therapy, unless considered stable by the treating investigator.
* Adequate venous access.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Step 2 Eligibility Confirmation

  * The following criteria must be confirmed within 7 days prior to lymphodepletion. If all criteria are not met, lymphodepletion should be delayed.

    * Confirmation of successful CAR-T manufacturing.
    * No evidence or suspicion of an infection.
    * Serum Creatinine ≤ 2 x institutional upper limit of normal (ULN) or eGFR >30 ml/min/1.73m2
    * No worsening of clinical status compared to either the initial eligibility criteria that would, in the opinion of the treating physician, significantly increase the risk from lymphodepleting chemotherapy or exclude them from treatment with study CAR-T therapy.
* Step 3 Eligibility Confirmation

  * The following criteria must be confirmed prior to CAR-T therapy. If all criteria are not met, CAR-T therapy should be delayed.

    * No worsening of clinical status compared to either the initial eligibility criteria that would, in the opinion of the treating physician, significantly increase the risks from treatment with CAR-T therapy.
    * Confirmation that washout periods outlined in section 6.6 and Appendix 10 have been followed.

Exclusion Criteria:

* Autologous or allogeneic stem cell transplant or CAR-T therapy within 6 weeks of planned CAR-T cell infusion.
* Subjects with active infection that requires systemic treatment
* History of autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of immunosuppressive medication within 6 months.
* Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of child bearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.
* Receiving other investigational agents.
* Confirmation that washout periods listed in Appendix 10 have been followed.
* Major surgery 4 weeks prior to starting study drug or who have not fully recovered from major surgery.
* The diagnosis of another malignancy within ≤ 2 years before study enrollment, except for those considered to be adequately treated with no evidence of disease or symptoms and/or will not require therapy during the study duration (i.e., basal cell or squamous cell skin cancer, carcinoma in situ of the breast, bladder or of the cervix, or low-grade prostate cancer with Gleason Score ≤ 6). Patients with transformed disease are allowed.
* Known brain metastases or cranial epidural disease. Note: Brain metastases or cranial epidural disease adequately treated with radiotherapy and/or surgery and stable for at least 4 weeks before the first dose of study treatment will be allowed on trial. Subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the first dose of study treatment.
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class III or IV, unstable angina pectoris, serious cardiac arrhythmias.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 3 months before the first dose.
    * QTc prolongation defined as a QTcF > 500 ms.
    * Known congenital long QT.
    * Left ventricular ejection fraction < 55%.
    * Uncontrolled hypertension defined as ≥ 140/90 as assessed from the mean of three consecutive blood pressure measurements taken over 10 minutes.
  * Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [subjects may not receive the drug through a feeding tube], social/ psychological issues, etc.)
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or seropositive HIV. Note: Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity to investigational product (IP) or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.6 and Appendix 10. Unless otherwise stated, a washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.
* Subjects with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Production and infusion of CAR-T therapy in 5/6 patients who have undergone successful apheresis and no more than 3/6 patients with ≥ grade 3 non-hematological CAR-T related toxicities or events of special interest within 28 days of CAR-T administration. | 28 days
  To assess the feasibility of administering CAR-T cells targeting CD19 for the treatment of relapsed/refractory B cell lymphomas, relapsed/refractory chronic lymphocytic leukemia (CLL), Richter's Syndrome, or relapsed/refractory acute lymphoblastic leukemia (ALL). Feasibility is defined as production and infusion of CAR-T therapy in 5/6 patients who have undergone successful apheresis and no more than 3/6 patients with ≥ grade 3 non-hematological CAR-T related toxicities or Events of Special Interest within 28 days of CAR-T administration.

SECONDARY OUTCOMES:
Objective response rate (ORR) defined as the proportion of subjects achieving a confirmed PR or CR at Day 28 and Month 3. | 3 months
  To assess the objective response rates (ORR) of subjects who have received anti-CD19 CAR-T cells
Disease free survival at 1 year post CAR-T administration based on 2014 Lugano Criteria (NHL patients) , IWCLL criteria (CLL patients) or EWALL recommendations (ALL patients). | 1 year
  To assess disease-free survival (DFS)
Overall survival as defined as the time from CAR-T administration until 6 months and 12 months post CAR-T administration | 12 months
  To assess overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Patel, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States